CLINICAL TRIAL: NCT07403266
Title: Treatment With Full-spectrum Cannabis Extract of Refractory Epilepsy Associated With Tuberous Sclerosis Complex (TSC)
Acronym: Spectrum
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oils4Cure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EstuEla2022; 2024-520171-27-00 (EU CTIS Number)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Tuberous Sclerosis Complex (TSC)
Keywords: Refractary Epilepsy
MeSH Terms: conditions — Tuberous Sclerosis

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind clinical trial with two treatment arms, randomized 1:1, placebo-controlled (part 1), followed by an open-label phase with a single treatment arm using the investigational product (part 2).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Randomized patients assigned to the active treatment group.
  Interventions: Drug: YCJ-01 Full Spectrum cannbis Extract
- placebo (Placebo Comparator): Randomized patients assigned to the placebo group.
  Interventions: Drug: YCJ-01 Full Spectrum cannbis Extract; Drug: Placebo

INTERVENTIONS:
Drug: YCJ-01 Full Spectrum cannbis Extract — Ful Spectrum cannabis extract
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
1. To assess treatment efficacy with YCJ-01 by changes in the number of epileptic seizures in patients with refractory epilepsy secondary to Tuberous Sclerosis Complex. 2. To assess the safety of the treatment with YCJ-01 in patients with refractory epilepsy secondary to Tuberous Sclerosis Complex.

DETAILED DESCRIPTION:
The current situation of epilepsy is a very frequent problem with onset in the first years of life in patients with tuberous sclerosis complex (TSC). There are many current therapeutic options; however, 63.3% of patients have uncontrolled epilepsy and most of them experience daily seizures. Poor seizure control is correlated with intellectual disability and autism spectrum disorder. Given the lack of effective treatments for the management of refractory epilepsy, a prospective, experimental clinical trial has been designed. Although there are additional treatment options such as vagus nerve stimulation and the ketogenic diet (apart from antiepileptic drugs), they do not control epilepsy.

Comparison of the number of monthly seizures since the initiation of the treatment with YCJ-01 with respect to the baseline period: in patients assigned to receive YCJ-01, change in the number of monthly seizures in the second month of treatment with respect to the baseline period; and in patient assigned to receive a placebo, changes in the number of monthly seizures in the second month of treatment with YCJ-01 with respect to the baseline period.

Occurrence of Adverse Events (AE), Severe AE (SAE), AE resulting in study treatment withdrawal, AE of special interest (AESI), and changes in vital signs and laboratory values during the clinical trial. (Variable associated to the primary objective 2). To assess the response rate to YCJ-01/placebo: patients who achieve a decrease in at least a 50 % of the number of epileptic seizures compared to the baseline period (from visit P0 to P1) will be considered responders.

To assess the proportion of subjects in treatment with YCJ- 01/placebo who achieve a 25%, 50%, 75%, or 90% reduction compared to the baseline period (from visit P0 to P1) in the number of epileptic seizures To assess the proportion of patients in treatment with YCJ-01/placebo free of seizures since the initiation of the assigned treatment.

To assess the effect of YCJ-01 on control of epileptic seizures (changes in seizure severity and types) before and after the initiation of the treatment.

Comparison of the number of monthly epileptic seizures between the two treatment groups and the baseline period: change in number of monthly seizures of patients assigned to receive the investigational medicinal product during the second month of treatment (from visit P2 to P3) with respect of the baseline period (from visit P0 to P1), in comparison to the second month of treatment (from visit P2 to P3) to the group receiving placebo with respect to the baseline period (from visit P0 to P1).

Comparison of the number of monthly seizures since the initiation of the treatment with YCJ-01 with respect to the baseline period: in patients assigned to receive YCJ-01, change in the number of monthly seizures in the months of treatment after the second month of treatment with respect to the baseline period; and in patients assigned to receive placebo, changes in the number of monthly seizures in the months of treatment after the second month of treatment with YCJ-01 with respect to baseline Comparison of the number of monthly seizures once the final dose was reached in P4-P5 with respect to the baseline period (from visit P0 to P1) in each of the patients. (Variable associated with primary objective 1).

Response rate to YCJ-01: patients who achieve a decrease of at least a 50 % of the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) in visits P3, P4, P6, and P7 will be considered responders. (Variable associated to the secondary objective 1).

Response rate to YCJ-01in comparison to the placebo group: patients who achieve a decrease in at least a 50 % of the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) in visit P3 will be considered responders. (Variable associated to the secondary objective 1).

Proportion of subjects in treatment with YCJ-01 achieving a 25%, 50%, 75%, 90% reduction in the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) at visits P3, P4, P6, and P7. (Variable associated to the secondary objective 2).

Proportion of subjects in treatment with YCJ-01 compared to placebo group achieving a 25%, 50%, 75%, 90% reduction in the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) at visit P3. (Variable associated to the secondary objective 2).

Proportion of patients in treatment with YCJ-01 free of epileptic seizures: defined as those participants with no seizure of any type from the initiation of the treatment with YCJ-01 till visit P7, or a period of time that doubles the baseline maximum interval between seizures (International League Against Epilepsy, ILAE). (Variable associated with the secondary objective 3).

Proportion of patients in treatment with YCJ-01 free of epileptic seizures in comparison to the placebo group: defined as those participants with no seizure of any type from the initiation of the assigned treatment till visit P7, or a period of time that doubles the baseline maximum interval between seizures (International League Against Epilepsy, ILAE). (Variable associated with the secondary objective 3).

Effect on control of epileptic seizures (variable associated to the secondary objective 4): Changes in severity and in types of epileptic seizures will be assessed after the initiation of the treatment (from visit P1 to P2, from visit P2 to P3, from visit P3 to P4, from visit P4 to P5, from visit P5 to P6, from visit P6 to P7) with respect to the baseline period (form visit P0 to P1).Comparison of the number of monthly epileptic seizures between the two treatment groups and the baseline period: change in number of monthly seizures of patients assigned to receive the investigational medicinal product during the second month of treatment (from visit P2 to P3) with respect of the baseline period (from visit P0 to P1), in comparison to the second month of treatment (from visit P2 to P3) to the group receiving placebo with respect to the baseline period (from visit P0 to P1).

Comparison of the number of monthly seizures since the initiation of the treatment with YCJ-01 with respect to the baseline period: in patients assigned to receive YCJ-01, change in the number of monthly seizures in the months of treatment after the second month of treatment with respect to the baseline period; and in patients assigned to receive placebo, changes in the number of monthly seizures in the months of treatment after the second month of treatment with YCJ-01 with respect to baseline Comparison of the number of monthly seizures once the final dose was reached in P4-P5 with respect to the baseline period (from visit P0 to P1) in each of the patients. (Variable associated with primary objective 1).

Response rate to YCJ-01: patients who achieve a decrease of at least a 50 % of the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) in visits P3, P4, P6, and P7 will be considered responders. (Variable associated to the secondary objective 1).

Response rate to YCJ-01in comparison to the placebo group: patients who achieve a decrease in at least a 50 % of the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) in visit P3 will be considered responders. (Variable associated to the secondary objective 1).

Proportion of subjects in treatment with YCJ-01 achieving a 25%, 50%, 75%, 90% reduction in the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) at visits P3, P4, P6, and P7. (Variable associated to the secondary objective 2).

Proportion of subjects in treatment with YCJ-01 compared to placebo group achieving a 25%, 50%, 75%, 90% reduction in the number of epileptic seizures with respect to the baseline period (from visit P0 to P1) at visit P3. (Variable associated to the secondary objective 2).

Proportion of patients in treatment with YCJ-01 free of epileptic seizures: defined as those participants with no seizure of any type from the initiation of the treatment with YCJ-01 till visit P7, or a period of time that doubles the baseline maximum interval between seizures (International League Against Epilepsy, ILAE). (Variable associated with the secondary objective 3).

Proportion of patients in treatment with YCJ-01 free of epileptic seizures in comparison to the placebo group: defined as those participants with no seizure of any type from the initiation of the assigned treatment till visit P7, or a period of time that doubles the baseline maximum interval between seizures (International League Against Epilepsy, ILAE). (Variable associated with the secondary objective 3).

Effect on control of epileptic seizures (variable associated to the secondary objective 4): Changes in severity and in types of epileptic seizures will be assessed after the initiation of the treatment (from visit P1 to P2, from visit P2 to P3, from visit P3 to P4, from visit P4 to P5, from visit P5 to P6, from visit P6 to P7) with respect to the baseline period (form visit P0 to P1).

ELIGIBILITY:
Inclusion Criteria:Patients of any sex between 2 and 65 years of age (both included) Diagnosis confirmed by the TSC investigator (by clinical criteria and/or genetic study).

Refractory epilepsy secondary to TSC, defined as that not responding successfully to traditional AEDs (2 or more), ketogenic diet, vagal nerve stimulator, and/or whose patients are not candidate for epilepsy surgery or persist with seizures after surgery.

Patients with a minimum of 4 epileptic seizures or more within 4 weeks prior to the initiation of the assigned treatment in the trial, with observable external signs (loss of consciousness or motor component).

Stability in AEDs doses, and in ketogenic diet/programming of the device associated with the vagal nerve stimulator with no changes for at least 4 weeks prior to the initiation of the assigned treatment.

Patients who are in treatment with 3 or less AEDs at the time of signing the informed consent. For the purposes of assessing eligibility, Clobazam will not be counted as AED Willingness by patients or caregivers/family members (in case of patients who are minors or under legal guardianship) to complete the seizure diary.

In case of women of child-bearing age, for safety, those who agree to follow the required contraceptive measures from the signing of the informed consent until three months after stop the intake of the investigational medicinal product.

Patients who have signed the informed consent either by themselves or through a legal representative.

-

Exclusion Criteria:Patients who are receiving treatment on corticoids at the time of signing the informed consent.

Pregnancy. Breastfeeding women To have participated in another clinical trial, unless at least 5 half- lives of the investigational product have elapsed, or 12 weeks, if it is a product with cannabis oil.

Patients who have received products with cannabis oil in the last 12 weeks. Patients who did not correctly follow the AED treatment in the 4 weeks prior to the intervention assigned in the trial.

Patients who changed medication or AED dose, ketogenic diet, or the vagal stimulator during the 4 weeks prior to the initiation of the intervention assigned in the trial.

Cardiac, renal, and hepatic failure, pancreatic insufficiency, or hematologic dysfunction with values above the normal limits of creatinine and urea; values 2 times the normal limits of transaminases, lipases, and serum amylase; platelets < 80000/mm3, and white blood cell count <3000/mm3.

Uncontrolled severe medical condition such as: hepatic disease, increased bilirubin levels more than twice the normal limit, cirrhosis, chronic hepatitis (hepatitis B or C), uncontrolled diabetes (defined as blood glucose >150 mg%), (chronic or acute) active infections or uncontrolled severe infections, or active bleeding.

Patients or family/caregivers (in case of patients who are minors or under legal guardianship) who does not agree to comply with the requirements and trial visits or present a high risk of non-compliance with the protocol, according to the treating physician.

Allergy to any of the components of the investigational medicinal product/placebo.

Family (considering only first-degree blood relatives) or personal history of schizophrenia.

Personal history of suicide attempts.

-

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
changes in the number of epileptic seizures in patients | 6 months
  1. To assess treatment efficacy with YCJ-01 by changes in the number of epileptic seizures in patients with refractory epilepsy secondary to Tuberous Sclerosis Complex. 2. To assess the safety of the treatment with YCJ-01 in patients with refractory epilepsy secondary to Tuberous Sclerosis Complex.
  Variables de Evaluación Primaria Comparison of the number of monthly seizures since the initiation of the treatment with YCJ-01 with respect to the baseline period: in patients assigned to receive YCJ-01, change in the number of monthly seizures in the second month of treatment with respect to the baseline period; and in patient assigned to receive a placebo, changes in the number of monthly seizures in the second month of treatment with YCJ-01 with respect to the baseline period.
  Occurrence of Adverse Events (AE), Severe AE (SAE), AE resulting in study treatment withdrawal, AE of special interest (AESI), and changes in vital signs and laboratory values during the clinical trial.

SECONDARY OUTCOMES:
To assess the response rate to YCJ-01/placebo | 6 months
  To evaluate the response rate to YCJ-01/placebo: responders will be defined as those patients who achieve at least a 50% reduction in the number of epileptic seizures compared with the baseline period (from visit P0 to P1).
  To evaluate the proportion of subjects treated with YCJ-01/placebo who achieve a 25%, 50%, 75%, or 90% reduction in the number of epileptic seizures compared with the baseline period (from visit P0 to P1).
  To evaluate the proportion of patients treated with YCJ-01/placebo who are seizure-free from the start of the assigned treatment.
  To evaluate the effect of YCJ-01 on seizure control (changes in seizure severity and types) before and after treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ruber Internacional, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: registro español de ensayos clínicos — https://reec.aemps.es/reec/estudio/2024-520171-27-00